CLINICAL TRIAL: NCT04843397
Title: PROspective Multicentre Study to Identify Diagnostic Key PERfOrmance Indicators in Upper GI Endoscopy (PROSPERO)
Brief Title: Diagnostic Performance Indicators in Upper GI Endoscopy:PROSPERO Study
Acronym: PROSPERO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Massimiliano di Pietro, MD, Senior Clinical Investigator Scientist, University of Cambridge
Other Study IDs: PROSPERO_protocol v1.0
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Esophageal Cancer; Gastric Cancer; Barrett Esophagus; Gastric Atrophy; Gastric Intestinal Metaplasia; Duodenal Adenoma; Esophageal Dysplasia; Duodenum Cancer; Gastric Polyp; Barretts Esophagus With Dysplasia
Keywords: upper GI endoscopy; esophagogastroduodenoscopy; esophageal cancer; gastric cancer; duodenal cancer; barretts esophagus; gastric polyp; premalignant upper GI lesions; upper GI cancer prevention; upper GI cancer early diagnosis; diagnostic upper GI endoscopy key performance indicators
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Barrett Esophagus; Gastritis, Atrophic; Duodenal Neoplasms; Polyposis, Gastric

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Clinical samples from biopsies taken during endoscopic procedures for the purpose of tissue diagnosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Arm: Patients referred for clinically indicated EGD, without known precancerous condition. Patients will receive endoscopy with standardised biopsy and photodocumentation protocol

SUMMARY:
Cancers of the upper gastro-intestinal tract, including esophagus (gullet), stomach and small bowel, are amongst the deadliest malignancies. The main reason for their high mortality rate is that they are usually diagnosed late when curative treatments are no longer effective. However, these types of cancer generally arise from well-described pre-cancerous diseases, such as Barrett's esophagus and gastric intestinal metaplasia. This provides an opportunity for clinicians to detect these pre-cancerous conditions early and offer adequate cure or clinical monitoring before they progress to cancer. A camera test (gastroscopy) is the gold-standard test to detect pre-cancerous diseases in these organs.

There has been limited research to set the standards for performance of a gastroscopy, especially with regards to diagnosis of pre-cancerous conditions, which require knowledge and skills by the physician performing the test (endoscopist). Therefore, the hypothesis behind this study is that the aforementioned pre-cancerous diseases are understudied and often go undetected. This study aims to understand how often endoscopists should diagnose these pre-cancerous diseases on routine gastroscopy and help define the standards to measure performance. The investigators will assess the following rates: i. how often endoscopists diagnose these pre-cancerous lesions during endoscopy; ii. How often these conditions are diagnosed on biopsies taken according to a standardized protocol; iii. How often these condition should have been diagnosed by the endoscopists based on the review of pictures by expert endoscopists. The investigators will also compare the rates of correct diagnosis by endoscopists with different levels of experience and based on the times spent to complete the diagnostic test.

Investigating these aspects will enhance the understanding of the medical community with regards to the diagnosis of these pre-cancerous lesions and set endoscopy standards to improve their early detection and treatment before they progress to cancer. This will translate to improved cancer prevention and benefit for patients.

DETAILED DESCRIPTION:
BACKGROUND Esophagogastroduodenoscopy (EGD) is the gold-standard test for investigating upper gastrointestinal (GI) tract pathology. The learning curve for EGD is generally steep and it is often performed by trainees at the mid stages of core training as well as nurse endoscopists. Currently the Joint Advisory Group for GI endoscopy (JAG) recommends a minimum number of 200 procedures to acquire the skills and perform endoscopy independently. However, there has been very little research done to set the standard required to measure EGD performance. The only validated quality indicators in EGD include the successful J-manoeuvre rate and D2 intubation rate, which reflect very basic skills and do not measure diagnostic ability. This contrasts with key performance indicators (KPI) for colonoscopy, for which extensive research has led to development of formal quality performance indicators. In colonoscopy formal quality indicators include (i) cecal intubation rate, (ii) adenoma detection rate, (iii) rectal retroversion rate, (iv) colonoscopy withdrawal time, (v) polyp retrieval rate, (vi) post-colonoscopy colorectal cancer rate and (vii) perforation rate. This has allowed researchers to demonstrate that poor quality colonoscopy leads to an increase in the incidence of interval cancers.

Similar benchmarks have not been set for the upper GI tract. A recent UK study revealed that 7.7% cases of upper GI cancers were missed on previous EGD and that there was a correlation between missed cancer and high number of procedures per lists and hence, arguably, those performed under user time pressure. This is in line with studies on other Western populations indicating that between 5.3% and 13.9% of patients with upper GI cancers have had normal EGD reported within the previous 3 years. Given that gastroscopy is the most commonly performed procedure in endoscopy units in the UK and its demand is increasing, there is an urge to identify diagnostic KPI to measure diagnostic skills, to improve quality of the endoscopies and to reduce the rate of missed diagnoses. Furthermore, such minimum quality standards are extremely important to counteract the potential negative effects on the performance of the pressure faced by endoscopy departments to deliver diagnostic and therapeutic procedures in a timely fashion. The importance of adequate procedure time for diagnostic accuracy has been demonstrated both in the detection of oesophageal and gastric neoplastic lesions. For detection of upper GI neoplasia, it has been demonstrated that a minimum of 7 minutes per procedure should be spent in order to ensure adequate visualisation and allow detection of high-risk lesion . In a Korean study, that compared faster with slower endoscopists, all of whom had adequate training and experience, the slower endoscopists (withdrawal time from duodenum >3min) had a significantly higher detection rate of upper GI neoplasia. Finally, in the context of Barrett's oesophagus (BO), longer inspection times during EGD correlated with increase detection rate.

Pre-malignant lesions in the upper GI tract are generally understudied when compared to those in the lower GI tract. Furthermore, their epidemiology seems to vary with geography, and this has not been inadequately investigated in the UK. Barrett's esophagus (BE) is the only known precursor to esophageal adenocarcinoma. The population prevalence is difficult to estimate given that the condition can be asymptomatic, and the diagnosis is only made by endoscopy and biopsy. It is estimated that the prevalence in the general population in Western Countries is 1-2% with significant geographic variation, but increases in patients undergoing endoscopic procedures (4.0% in Dutch population, 5.6% USA). However, the majority of studies looking at BE prevalence are confounded by the fact that most procedures were performed for GERD symptoms generating selection bias. In studies performed in patients referred for colonoscopy (n=1500 approximately) the prevalence of BE varied between 6.8% and 16.7%.

Similar to oesophageal cancer, gastric cancer has its own pre-malignant precursors including gastric intestinal metaplasia (GIM) and gastric atrophy (GA) . The endoscopic diagnosis of GA and GIM however is not straightforward as the colorimetric shift from normal to pathological mucosa is subtle and additional endoscopic signs such as disappearance of gastric folds can be affected by the degree of air insufflation. The prevalence of GA can reach up to 33.3% in Western Europeans and is higher in East Asia. For GIM, the reported population prevalence in Western Countries ranges from 7 to 28.6%. These rates are however probably affected by selection bias, such as enrichment of individuals affected by H. pylori infection. In a Dutch study on patient referred for colonoscopy 0.8% had GA, 7.1% had both GA and GIM and 1.4% had gastric dysplasia.

For esophageal squamous dysplasia, the precursor lesion of oesophageal squamous cell carcinoma, prevalence estimates are between 3 and 38%. This reflects the variation in endoscopic methods, histopathological scoring and the studied populations from high-risk geographic regions such has Korea. The prevalence of squamous dysplasia in Western Countries in not well known, since it is generally very difficult to diagnose on white light endoscopy. It can be argued that squamous dysplasia is vastly underdiagnosed in clinical practice as the ratio between oesophageal adenocarcinoma and squamous cell carcinoma in the UK is just over 2:1, however squamous dysplasia is rarely diagnosed.

Duodenal adenoma is another understudied pre-malignant lesion that can in fact undergo malignant transformation in 30-85% of cases and as such, needs to be recognised and treated early and definitively . These occur very often in the context of familial adenomatous polyposis (FAP) syndrome, whereas sporadic duodenal adenomas are much rarer with a prevalence of 0.03-0.4% (32, 33).

The majority of studies looking at prevalence of pre-malignant upper GI conditions in the general population referred for EGD are limited by the lack of standardised endoscopy and biopsy protocols. In addition, none of the studies looked at variation of prevalence based on experience. Furthermore, no expert review of endoscopic images has been performed to ensure quality of the diagnosis. Although quality standards in upper GI endoscopy have been proposed by the British Society of Gastroenterology and European Society of Gastrointestinal Endoscopy, the majority of the statements in these guidelines have a low level of evidence and weak to moderate strength of the recommendation. Most importantly, none of the statements refer to diagnostic KPI, given that the expected detection rate of the upper GI pre-neoplastic and early neoplastic lesions at endoscopy is unknown. This represents a gap that our study aims to tackle.

HYPOTHESIS The hypothesis is that the prevalence of upper Gi pre-malignant condition is underestimated based on available literature data and that the detection rate of pre-cancerous upper GI lesions improves with a more rigorous and systematic approach to performing EGD. In the future, using diagnostic KPI to monitor performance of upper GI endoscopists will result in improved outcomes of oesophago-gastric cancer.

STUDY OBJECTIVES The aim of this study is to assess endoscopic and pathological outcomes during routine EGD using standard photo-documentation and biopsy protocol.

The primary objective is to define the prevalence of pre-malignant or early malignant upper GI tract lesions as measured by a standardised endoscopy and biopsy protocol. This is further broken down into categories of pre-malignant pathology, namely: 1) Barrett's esophagus with and without dysplasia; 2) squamous dysplasia;, 3) gastric atrophy/gastric intestinal metaplasia; , 4) gastric adenoma; and 5) duodenal adenoma.

The secondary objectives are:

1. Missed rate of endoscopic diagnosis compared to pathological diagnosis
2. Missed rate of endoscopic diagnosis compared to expert review of endoscopic photos
3. Correlation between duration of the endoscopy and detection of pre-neoplastic and neoplastic lesions
4. Quality of the endoscopic pictures taken in routine endoscopy
5. Correlation between endoscopist experience and rate of detection
6. Correlation between use of image enhanced endoscopy and rate of detection
7. Interobserver agreement among expert and not expert endoscopists
8. Correlation between life-style factors and pathological outcomes

STUDY DESIGN This will be a multicenter population study. Recruiting centers will be a range of Teaching and District General Hospitals in England. 1000 patients referred for urgent or routine endoscopy to evaluate upper GI symptoms will be recruited. The detection rates of upper GI tract pre-malignant lesions in our study procedures will be compared to standard historical data from each participating institution. An equivalent population from the year prior to the start of recruitment, matched for age, sex, indication for endoscopy and referral pathway, will be retrieved from the archives of each participating NHS Trust and directly contrasted to this study population to evaluate whether the detection rate of pre-malignant upper GI tract lesions improves with a more rigorous and systematic approach to performing EGD using a standardized photo documentation and biopsy protocol. In this way, the investigators can evaluate the immediate impact of our study and the utility of the proposed diagnostic KPI. As an example, the investigators already have date to show that in 2019 over 8,500 EGD were performed in Cambridge alone, of which 53% had biopsies taken. Based on matched pathology record, only 29 new diagnoses of GA or GIM were made during the same time period, suggesting the possibility of large under-detection of premalignant stomach. The endoscopic pictures will be evaluated by two expert endoscopists with interest in detection and treatment of upper GI pre-malignant and early malignant conditions. The quality of the pictures will be scored on a visual analogue scale based on two parameters: optical quality and representation of the intended section of the upper GI tract. The endoscopists will note the presence of premalignant conditions. In case of disagreement, a third investigator will review the picture to achieve a gold standard endoscopic diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, comprehend, and complete the consent form
2. Aged ≥18
3. Clinically fit for endoscopy
4. Referred for endoscopy via any clinical pathway

Exclusion Criteria:

1. Known upper GI conditions with or without ongoing endoscopic monitoring including Barrett's oesophagus, oesophageal dysplasia, gastric ulcers, duodenal polyps or any established upper GI malignancy
2. Previous oesophagectomy, gastrectomy for malignant disease
3. OGD performed within last 3 years of study initiation
4. Oesophageal stricture precluding completion of diagnostic endoscopic examination
5. Coagulopathy or anticoagulant/antiplatelet therapy for high risk conditions making non possible to discontinue the medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient referred and clinically fit for endoscopy via any clinical referral pathway that is able to consent to study participation.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Define the prevalence of pre-malignant upper GI tract lesions as measured by standardised endoscopy and biopsy protocol | 1 year
  The primary outcome is calculating the proportion of patients diagnosed with pre-malignant pathology in the upper GI tract. This is further broken down into categories of pre-malignant pathology, namely; 1) duodenal adenoma, 2) gastric atrophy/gastric intestinal metaplasia (IM), 3) gastric adenoma, 4) Barrett's oesophagus and 5) squamous dysplasia.
  The detection rates of upper GI tract pre-malignant lesions in our study procedures will be compared to standard historical data currently available to update and guide future practice guidelines.

SECONDARY OUTCOMES:
Missed rate of endoscopic diagnosis compared to pathological diagnosis | 1 year
  (defined as any pathological diagnosis that was not suspected by the endoscopist on visualisation alone)
Missed rate of endoscopic diagnosis compared to expert review of endoscopic photos | 1 year
  (defined as endoscopic lesions identified by expert review and not reported by primary endoscopist)
Correlation between duration of the endoscopy and detection of pre-neoplastic and neoplastic lesions | 1 year
  Assessment of whether duration of the endoscopy associates with diagnosis of pre-neoplastic lesions
Quality of the endoscopic pictures taken in routine endoscopy | 1 year
  defined as quantitative assessment of photo on a Visual Analogue Scale by expert endoscopists
Correlation between prevalence of diagnoses and endoscopist experience | 1 year
  Assessment of whether year of endoscopy practice correlate with the rate of detection of pre-malignant lesions
Correlation between use of image enhanced endoscopy and rate of detection | 1 year
  Assessment of whether use of dye or electronic chromoendoscopy improves detection of lesions
Interobserver agreement among expert and not expert endoscopists | 1 year
  Agreement will be assess with Cohen kappa values
Correlation between life-style factors and pathological outcomes | 1 year
  Assessment of utility of life-style information to predict diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Di Pietro, MD, Study Chair — MRC Cancer Unit,Hutchison/MRC Research Centre; Ines Modolell, MD, Principal Investigator — Cambridge University Hospitals; Andreas V Hadjinicolaou, Principal Investigator — Cambridge University Hospitals

REFERENCES:
- [Background] Rees CJ, Thomas Gibson S, Rutter MD, Baragwanath P, Pullan R, Feeney M, Haslam N; British Society of Gastroenterology, the Joint Advisory Group on GI Endoscopy, the Association of Coloproctology of Great Britain and Ireland. UK key performance indicators and quality assurance standards for colonoscopy. Gut. 2016 Dec;65(12):1923-1929. doi: 10.1136/gutjnl-2016-312044. Epub 2016 Aug 16. PMID 27531829
- [Background] Kaminski MF, Regula J, Kraszewska E, Polkowski M, Wojciechowska U, Didkowska J, Zwierko M, Rupinski M, Nowacki MP, Butruk E. Quality indicators for colonoscopy and the risk of interval cancer. N Engl J Med. 2010 May 13;362(19):1795-803. doi: 10.1056/NEJMoa0907667. PMID 20463339
- [Background] Tai FWD, Wray N, Sidhu R, Hopper A, McAlindon M. Factors associated with oesophagogastric cancers missed by gastroscopy: a case-control study. Frontline Gastroenterol. 2019 Jul 11;11(3):194-201. doi: 10.1136/flgastro-2019-101217. eCollection 2020. PMID 32419910
- [Background] Teh JL, Tan JR, Lau LJ, Saxena N, Salim A, Tay A, Shabbir A, Chung S, Hartman M, So JB. Longer examination time improves detection of gastric cancer during diagnostic upper gastrointestinal endoscopy. Clin Gastroenterol Hepatol. 2015 Mar;13(3):480-487.e2. doi: 10.1016/j.cgh.2014.07.059. Epub 2014 Aug 10. PMID 25117772
- [Background] Park JM, Huo SM, Lee HH, Lee BI, Song HJ, Choi MG. Longer Observation Time Increases Proportion of Neoplasms Detected by Esophagogastroduodenoscopy. Gastroenterology. 2017 Aug;153(2):460-469.e1. doi: 10.1053/j.gastro.2017.05.009. Epub 2017 May 10. PMID 28501581
- [Background] Gupta N, Gaddam S, Wani SB, Bansal A, Rastogi A, Sharma P. Longer inspection time is associated with increased detection of high-grade dysplasia and esophageal adenocarcinoma in Barrett's esophagus. Gastrointest Endosc. 2012 Sep;76(3):531-8. doi: 10.1016/j.gie.2012.04.470. Epub 2012 Jun 23. PMID 22732877
- [Background] Gerson LB, Shetler K, Triadafilopoulos G. Prevalence of Barrett's esophagus in asymptomatic individuals. Gastroenterology. 2002 Aug;123(2):461-7. doi: 10.1053/gast.2002.34748. PMID 12145799
- [Background] Hirota WK, Loughney TM, Lazas DJ, Maydonovitch CL, Rholl V, Wong RK. Specialized intestinal metaplasia, dysplasia, and cancer of the esophagus and esophagogastric junction: prevalence and clinical data. Gastroenterology. 1999 Feb;116(2):277-85. doi: 10.1016/s0016-5085(99)70123-x. PMID 9922307
- [Background] Ronkainen J, Aro P, Storskrubb T, Johansson SE, Lind T, Bolling-Sternevald E, Vieth M, Stolte M, Talley NJ, Agreus L. Prevalence of Barrett's esophagus in the general population: an endoscopic study. Gastroenterology. 2005 Dec;129(6):1825-31. doi: 10.1053/j.gastro.2005.08.053. PMID 16344051
- [Background] Joo YE, Park HK, Myung DS, Baik GH, Shin JE, Seo GS, Kim GH, Kim HU, Kim HY, Cho SI, Kim N. Prevalence and risk factors of atrophic gastritis and intestinal metaplasia: a nationwide multicenter prospective study in Korea. Gut Liver. 2013 May;7(3):303-10. doi: 10.5009/gnl.2013.7.3.303. Epub 2013 May 13. PMID 23710311
- [Background] Petersson F, Borch K, Franzen LE. Prevalence of subtypes of intestinal metaplasia in the general population and in patients with autoimmune chronic atrophic gastritis. Scand J Gastroenterol. 2002 Mar;37(3):262-6. doi: 10.1080/003655202317284156. PMID 11916187
- [Background] Kim N, Park YS, Cho SI, Lee HS, Choe G, Kim IW, Won YD, Park JH, Kim JS, Jung HC, Song IS. Prevalence and risk factors of atrophic gastritis and intestinal metaplasia in a Korean population without significant gastroduodenal disease. Helicobacter. 2008 Aug;13(4):245-55. doi: 10.1111/j.1523-5378.2008.00604.x. PMID 18665932
- [Background] den Hoed CM, van Eijck BC, Capelle LG, van Dekken H, Biermann K, Siersema PD, Kuipers EJ. The prevalence of premalignant gastric lesions in asymptomatic patients: predicting the future incidence of gastric cancer. Eur J Cancer. 2011 May;47(8):1211-8. doi: 10.1016/j.ejca.2010.12.012. Epub 2011 Jan 14. PMID 21239166
- [Background] Taylor PR, Abnet CC, Dawsey SM. Squamous dysplasia--the precursor lesion for esophageal squamous cell carcinoma. Cancer Epidemiol Biomarkers Prev. 2013 Apr;22(4):540-52. doi: 10.1158/1055-9965.EPI-12-1347. PMID 23549398
- [Background] Jepsen JM, Persson M, Jakobsen NO, Christiansen T, Skoubo-Kristensen E, Funch-Jensen P, Kruse A, Thommesen P. Prospective study of prevalence and endoscopic and histopathologic characteristics of duodenal polyps in patients submitted to upper endoscopy. Scand J Gastroenterol. 1994 Jun;29(6):483-7. doi: 10.3109/00365529409092458. PMID 8079103
- [Background] Beg S, Ragunath K, Wyman A, Banks M, Trudgill N, Pritchard DM, Riley S, Anderson J, Griffiths H, Bhandari P, Kaye P, Veitch A. Quality standards in upper gastrointestinal endoscopy: a position statement of the British Society of Gastroenterology (BSG) and Association of Upper Gastrointestinal Surgeons of Great Britain and Ireland (AUGIS). Gut. 2017 Nov;66(11):1886-1899. doi: 10.1136/gutjnl-2017-314109. Epub 2017 Aug 18. PMID 28821598